CLINICAL TRIAL: NCT05711693
Title: Integrated Silicon Photonics for Cardiovascular Disease Monitoring InSiDe-CC Clinical Validation of the Diagnostic Device (LDV) for the Measurement of Heart-carotid Pulse Wave Velocity (PWV) by Magnetic Resonance Imaging (MRI)
Brief Title: Measurement of Heart-carotid Pulse Wave Velocity (hcPWV) by Laser Doppler Vibrometry (LDV)
Acronym: InSide-CC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: C21-28; 2021-A02896-35 (Registry Identifier: IDRCB)
Record Dates: First submitted 2023-01-06; First posted 2023-02-03 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2024-11

CONDITIONS: Hypertension; Aortic Aneurysm; Bicuspid Aortic Valve; Marfan Syndrome; Aortic Dilatation
Keywords: stiffness; hypertension; ascending aorta
MeSH Terms: conditions — Hypertension; Aortic Aneurysm; Bicuspid Aortic Valve Disease; Marfan Syndrome | interventions — Blood Pressure; Heart Rate

STUDY DESIGN:
Intervention Model Description: Comparison of methods
Masking Description: MRI doctors will be blinded concerning LDV PWV values. Doctors performing LDV will not have access to MRI reports. Data will be consolidated and database frozen before reconciling MRI and LDV data
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Technique comparison (Experimental): All patients will undergo successively LDV heart to carotid PWV and ascending aorta PWV by MRI, for comparison
  Interventions: Device: Laser doppler vibrometry (LDV), heart(cordium) carotid pulse wave velocity (ccPWV); Procedure: Blood pressure and heart rate measurement; Device: carotid to femoral PWW measurement; Procedure: Questionnaire completion

INTERVENTIONS:
Device: Laser doppler vibrometry (LDV), heart(cordium) carotid pulse wave velocity (ccPWV) — Patients scheduled for thoracic aorta MRI will have LDV measurement of ccPWV. Both techniques will be compared
Procedure: Blood pressure and heart rate measurement — To all patients:
  - blood pressure and heart rate will be measured
Device: carotid to femoral PWW measurement — To all patients:
  - carotid to femoral PWW will be measured by LDV and tonometry for comparison
Procedure: Questionnaire completion — All patients will complete a questionnaire of acceptability

SUMMARY:
Aortic stiffness is an important imaging biomarker of vascular aging. The ascending aorta is the most elastic segment, and it is excluded by reference non-invasive method carotid to femoral pulse wave velocity (PWV). We propose to use laser-doppler vibrometry (LDV) to record superficial vibrations generated by cardiac activity and arterial pulses for measuring heart carotid PWV, a surrogate for ascending aorta.

The trial aims to demonstrate the equivalence between heart-carotid PWV made by laser-doppler vibrometry (LDV) with the reference MRI measurement (4D-FLOW MRI).

As secondary objectives, A) we aim to assess the reproducibility of LDV, compared with MRI, B) show that aortic stiffness measured by LDV fulfils international recommendations, C) to study the association between PWV and age or other cardiovascular risk factors, D) assess the acceptability of the measurement. For this, we include 100 consecutive patients, 50 women, 50 men, scheduled for clinically indicated thoracic aorta MRI.

DETAILED DESCRIPTION:
Cardiovascular (CV) diseases and their risk factors are the leading causes of morbidity and mortality in the world. They are responsible for more than 17.3 million deaths per year worldwide, accounting for 30% of all causes of death.

The measurement of arterial stiffness is useful to estimate the global CV risk with more precision than the simple point assessment of the classical cardiovascular risk factors.

Carotid-femoral pulse wave velocity (cfPWV) by tonometry is the reference method. However, it excludes by principle the ascending aorta, which is the most distensible and physiologically the most important segment. The InSiDe project aims to measure heart - carotid pulse wave velocity (hcPWV) from the measurement of skin vibrations on the chest and neck by laser doppler vibrometry (LDV), enclosing principally the ascending aorta. This will allow the measurement and validation of a new biomarker that quantifies the stiffness of the ascending aorta. We have demonstrated a very good agreement of the LDV-based cfPWV with the reference technique by tonometry. Our hypothesis, based on physiological reasons, is that heart-carotid PWV will surpass carotid-femoral PWV as a biomarker of large artery stiffness.

The trial aims to demonstrate the equivalence between heart-carotid PWV measured by laser-doppler vibrometry (LDV) with the reference MRI measurement (4D-FLOW MRI). MRI, the gold standard comparator is technically demanding and uncomfortable for the patient, much more expensive and not applicable at the general population level. It is therefore likely that measurement by laser-doppler vibrometry, without contact, more comfortable, acceptable and fast, could replace MRI for mass applications.

For this, we include 100 consecutive patients, 50 women, 50 men, scheduled for clinically indicated thoracic aorta MRI.

ENDPOINTS

Primary endpoint:

• Heart-carotid PWV measured by LDV. To evaluate the agreement between heart-carotid PWV measured by LDV and the same measurement made by MRI (plus 4D-FLOW MRI) of the thorax.

Secondary endpoints:

* Reproducibility of the LDV hcPWV
* Measurement of LDV cfPWV compared with tonometry
* Association between PWV (hc, cf, LDV, MRI), and age, other risk factors
* Assessment of patient acceptability of the measurement

Statistical analysis The statistical technique used will be the Bland - Altman plot and the corresponding bias assessment (mean Bland-Altman bias and limits of agreement, defined as the mean bias ±1.96 - standard deviation, are provided); the coefficient of variation (CV) will also be used.

Description of the device being investigated:

The LDV device, developed by the European consortium CARDIS (Medtronic,SIOS, iMEC, Tyndall Institute) uses two arrays with 6 laser beams. It is a non-invasive exploration, by category 1 laser without any risk for the patient and allows to measure the local arterial stiffness (to evaluate the heart-carotid PWV) and segmental without contact with the skin by using the LDV technique. In practice, this device allows the evaluation of the hcPWV from the measurement of skin vibrations on the chest and neck.

Description of the device used as a comparator:

The reference technique is MRI, used in combination with 4D-FLOW MRI, an innovative technique that allows full 3-dimensional anatomical coverage as well as velocity coding in all 3 directions, opening new and unique possibilities for visualizing and quantifying complex cardiovascular blood flow

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 90 years of age in both sexes, who visit the hospital for MRI thoracic MRI as part of routine care.
* Enrolled in a social security plan or beneficiary of such a plan.
* Free, informed, written consent signed by the participant and the investigator (no later than the day of inclusion and prior to any examination required by the research).

and before any examination required by the research and even before the thoracic MRI planned in the care setting).

Exclusion Criteria:

* Individuals under court protection, guardianship or under curator.
* MRI examination done in an emergency context
* Patients with skin lesions (severe eczema, wounds, etc.) in the thorax or neck that do not allow the application of not allowing the application of the skin protection film on the area of interest;
* Allergies to the adhesive film.
* Patients who have a beard, which would make it difficult to apply an adhesive cast.
* Subjects who are not affiliated with social security or an equivalent plan.
* Refusal or linguistic or psychic incapacity to read the information and not object to the research.
* Patients with a serious pathology threatening the vital prognosis in the short and medium term (cancer metastatic cancer, end-stage renal failure, end-stage liver failure, end-stage heart failure) heart failure).
* Patients with a history of acute severe (II, IV) heart failure.
* Patients with progressive cardiovascular pathologies (unstable coronary artery disease, severe valvular disease,stroke, aortic dissection).
* Rhythm disorders: atrial fibrillation, high degree auriculoventricular block.
* Pregnant or breastfeeding women
* Person subject to an exclusion period for another research

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-03-13 (Actual); Primary Completion 2024-06-19 (Actual); Study Completion 2024-06-19 (Actual)

PRIMARY OUTCOMES:
Heart-carotid pulse wave velocity (hcPWV) measured by LDV compared to MRI | 1 hour
  Values of PWV obtained by LDV and by MRI will be compared.

SECONDARY OUTCOMES:
Reproducibility of LDV heart-carotid pulse wave velocity (hcPWV) | 1 hour
  Measures will be duplicated and the average calculated, in case of discrepancy > 0.5 m/s, a third measurement is made and the median determined. Two series of measurements will be taken at 5minutes of interval.
Validity of carotid to femoral pulse wave velocity (cfPWV) measured by LDV | 1 hour
  Values of cfPWV obtained by LDV will be also compared with values obtained by tonometry.
Association of heart-carotid pulse wave velocity (hcPWV) measured by LDV with classical cardiovascular (CV) risk factors and disease | 1 hour
  The correlation coefficient and linear regression will be calculated.
Acceptability of heart-carotid pulse wave velocity (hcPWV) measured by LDV compared with MRI | 1 hour
  A questionnaire of acceptability will be completed by the patient after the measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Boutouyrie, Principal Investigator — Hôpital Européen Georges-Pompidou
Locations (1):
- Hôpital Européen Georges Pompidou, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beeckman S, Badhwar S, Li Y, Aasmul S, Madhu N, Khettab H, Mousseaux E, Gencer U, Boutouyrie P, Bruno RM, Segers P. Heart-carotid pulse-wave velocity via laser-Doppler vibrometry as a biomarker for arterial stiffening: a feasibility study. Physiol Meas. 2025 Apr 22;46(4). doi: 10.1088/1361-6579/adcb85. PMID 40209757